CLINICAL TRIAL: NCT07190625
Title: Intranasal Versus Intravenous Fentanyl For Procedural Analgesia in Preterm Neonates : A Randomized Controlled Trial
Brief Title: Intranasal Versus Intravenous Fentanyl For Procedural Analgesia in Preterm Neonates
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MD342/2023
Record Dates: First submitted 2025-09-05; First posted 2025-09-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Procedural Pain
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- intravenous group (Active Comparator): this group of neonates will recieve intravenous fentanyl during procedure
  Interventions: Drug: fentanyl intravenous
- direct intranasal group (Active Comparator): this group of neonates will recieve direct intranasal fentanyl during procedure
  Interventions: Drug: fentanyl intranasal direct
- nasal atomizer group (Active Comparator): this group of neonates will recieve intranasal fentanyl with atomizer during procedure
  Interventions: Drug: Fentanyl intranasal using atomizer

INTERVENTIONS:
Drug: fentanyl intravenous — giving intravenous fentanyl
  Arms: intravenous group
Drug: Fentanyl intranasal using atomizer — giving intranasal fentanyl using nasal atomizer
  Arms: nasal atomizer group
Drug: fentanyl intranasal direct — giving intranasal fentanyl directly into nostrils
  Arms: direct intranasal group

SUMMARY:
Pain in neonatal life has profound long-term developmental impacts, so pain control is crucial. The intranasal (IN) route is a minimally invasive method for rapidly delivering fentanyl to provide short-term analgesia and sedation in adults and pediatrics, but few data exist about its use in neonates. Meanwhile, intravenous fentanyl is widely used in sedation and pain management.

Using intranasal fentanyl as an analgesic in preterm neonates may provide a rapid, effective, noninvasive route for administration.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of intranasal fentanyl versus the intravenous route for procedural pain management in preterm neonates as assessed by pain scoring system before and after the procedure.

Enrolled neonates will be allocated randomly to one of the three groups during painful procedure, using single blinded method, as scoring will occur by a different physician than the researcher.

Atomizer group: will receive intranasal fentanyl (@fentanyl hamein 50 mcg/1 ml, manufactured by Sunny Pharmaceutical) using a nasal atomizer; the dose of INF is 1.5 µg/kg/dose.

Direct nasal group: will receive intranasal fentanyl directly installed into the nostrils with the same dose.

Typically, one dose is given during the procedure; after 5 minutes, a second dose could be administered based on the clinical assessment (maximum two doses per procedure), with reassessment of the pain score.

o Intravenous group: will receive intravenous fentanyl with a dose of 1 μg/kg as the standard of care.

All of the following data will be obtained:

Full history taking: antenatal, natal, and postnatal history Gestational age will be estimated using the date of the last menstrual period and confirmed by the new Ballard scoring system.

Full clinical examination: including general, cardiopulmonary, abdominal, and neurological examinations and anthropometric measurements.

Type of procedure done to the patient, number of attempts if more than once, and number of intranasal fentanyl doses needed.

Type of respiratory support at the time of intranasal fentanyl administration.

Effectiveness of intranasal fentanyl will be assessed using:

Premature Infant Pain Profile (PIPP) scale The pre-procedure PIPP scale will be recorded just before administration of the first dose of IN fentanyl and commencement of the painful procedure, while the post-procedure PIPP score will be recorded within 5 minutes of fentanyl administration.

PIPP scores range from 0 to 21. A PIPP score of 0-6 suggests minimal or no pain, 7-12 indicates moderate pain, and a score ≥ 13 is interpreted as severe pain.

Physiological parameters of heart rate, respiratory rate, oxygen saturation, blood pressure, and fraction of inspired oxygen (FiO2) at baseline (just before fentanyl administration) and at pre-specified intervals (15, 30, 45, and 60 min) after fentanyl use.

Monitor adverse events after fentanyl use, such as apnea (cessation of breathing for >20 s), bradycardia (heart rate < 100 beats/minute), desaturation (oxygen saturation < 80%) , and chest wall rigidity associated with laryngospasm for 60 min after IN fentanyl administration. Local effects include nasal discomfort and irritation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age between 28 and 36 weeks gestation.
* Undergoing painful procedures such as central venous access insertion, elective endotracheal intubation, and lumbar puncture.

Exclusion Criteria:

* known contraindications for fentanyl use, such as fentanyl hypersensitivity and liver failure.
* Known contraindication for intranasal administration of drugs (choanal atresia, nasal mucosal erosion, and epistaxis)
* Post-surgical patients.
* Patients sedated by fentanyl infusion / midazolam infusion.
* Evidence of neurological disease with disturbed conscious level, such as intraventricular hemorrhage grade III or IV, hypoxic ischemic encephalopathy, or inborn error of metabolism.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-12-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
procedural pain managment | from giving the fentanyl before the procedure till one hour after .
  The efficacy of different modalities of intranasal fentanyl, either nasal atomizer or direct method, versus intravenous administration in neonatal pain management using Premature Infant Pain Profile (PIPP) scale before and after the administration.
  PIPP score ranges from 0 to 21, A PIPP score of 0-6 suggests minimal or no pain, 7-12 indicates moderate pain and a score ≥ 13 is interpreted as severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Passant Fahmy, M.Sc, Principal Investigator — Assisstant lecturer
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided